CLINICAL TRIAL: NCT01389141
Title: Ovarian Follicular Wave Dynamics During The Menstrual Cycle: Relationship To Age, Reproductive Hormones And Musculoskeletal Health
Brief Title: Age-related Changes in Ovarian Follicular Wave Dynamics
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Foundation for Women's Health (Other)
Responsible Party: Principal Investigator, Angela Baerwald, M.D., University of Saskatchewan
Other Study IDs: RBRU-ARB 003
Record Dates: First submitted 2010-05-21; First posted 2011-07-07 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Aging
Keywords: ovary; follicle; hormones; bone; muscle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples are isolated and frozen for retrospective analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- mid-reproductive age
- late reproductive age-1
- late reproductive age-2

SUMMARY:
The investigators hypothesize that age-related changes in the number and growth dynamics of ovarian follicles will be associated with changes in hormone levels and corresponding changes in musculoskeletal health.

DETAILED DESCRIPTION:
The following hypotheses will be tested:

1. Differences in ovarian follicular wave dynamics will be detected in women of different ages;
2. The numbers and patterns of ovarian follicle waves in women are repeatable over multiple menstrual cycles;
3. Differences in inhibin B, inhibin A, and AMH will be detected in women with 2 versus 3 or more follicular waves
4. Differences in FSH, LH, progesterone, inhibin B, inhibin A, and AMH detected in MRA and LRA2 women, will change with the numbers of follicles and waves detected;
5. 'Luteal out of phase events' (aka LOOP cycles) will be more prevalent in LRA2 versus MRA women, and will represent major anovulatory waves and/or ovulatory waves;
6. When compared to MRA group, LRA2 women will have lower bone mineral mass and areal density at the lumbar spine; reduced trabecular density at the distal radius and thinner cortices with lower cortical density at the radial and tibial shaft. Other bone outcomes will be similar between the groups;
7. When compared to MRA group, LRA2 women will have lower total body lean mass, greater fat mass and less dense muscle tissue at the forearm and lower limb and lower hand grip strength.
8. Reduced bone mineral mass, areal density, trabecular density, cortical density and hand grip strength in LRA2 versus MRA women will be associated with reduced follicle number, a greater prevalence of LOOP cycles, higher serum FSH and lower inhibin concentrations

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Age of 18-55
* 18<BMI<35
* Menstrual cycle history:
* MRA group: regular cycles
* LRA-1 group: history of regular cycles, with variable cycles allowed (no more than 3 months amenorrhea)
* LRA-2 group: variable cycles allowed (no more than 3 months amenorrhea)
* Has not taken hormonal contraception within 2 months of initiating study procedures
* Agrees to use back-up contraception throughout the course of the study, if sexually active (condoms to be provided)
* 3.0 < Prolactin < 20.0 ug/L
* 0.30 < TSH < 5.50 mIU/L
* Normal complete blood count (CBC)
* Beta human Chorionic Gonadotropin < 5IU/L.

Exclusion Criteria:

* Smokers
* Documented ovarian failure
* History of or currently-diagnosed infertility of unexplained or female origin;
* Medical conditions known or suspected to interfere with reproductive function (including PCOS)
* Presence of only one ovary
* Ovaries inaccessible with transvaginal ultrasonography
* The use of any medications known or suspected to interfere with reproductive function
* Ongoing pregnancy
* Lactation
* Participation in an investigational drug trial in the 30 days prior to the pre-study visit
* Planning to undergo surgery during the course of the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Seventy healthy women, exhibiting all inclusion criteria and no exclusion criteria will be enrolled in this study. Women will be grouped into 1 of the following age categories:
  1. . Mid-reproductive age (MRA): 18-35 years
  2. . Late reproductive age-1 (LRA1): 36-44 years
  3. . Late reproductive age -2 (LRA2): 45-55 years (this group will include women in the LRA, EMT and LMT groups, as previously characterized by STRAW)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Follicle diameter (mm) | 4 years

SECONDARY OUTCOMES:
- Follicle number | 4 years
Serum FSH | 4 years
bone mineral density | 4 years
Serum LH | 4 years
Serum Estradiol | 4 years
Serum Progesterone | 4 years
Serum Inhibin A | 4 years
Serum Inhibin B | 4 years
Serum AMH | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Baerwald, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Reproductive Biology Research Unit, Department of Obstetrics, Gynecology and Reproductive Sciences, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. Characterization of ovarian follicular wave dynamics in women. Biol Reprod. 2003 Sep;69(3):1023-31. doi: 10.1095/biolreprod.103.017772. Epub 2003 May 14. PMID 12748128
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Derived] Bashir ST, Baerwald AR, Gastal MO, Pierson RA, Gastal EL. Follicle growth and endocrine dynamics in women with spontaneous luteinized unruptured follicles versus ovulation. Hum Reprod. 2018 Jun 1;33(6):1130-1140. doi: 10.1093/humrep/dey082. PMID 29659847
- [Derived] Baerwald A, Vanden Brink H, Hunter C, Beuker D, Lim H, Lee CH, Chizen D. Age-related changes in luteal dynamics: preliminary associations with antral follicular dynamics and hormone production during the human menstrual cycle. Menopause. 2018 Apr;25(4):399-407. doi: 10.1097/GME.0000000000001021. PMID 29112593
- [Derived] Vanden Brink H, Robertson DM, Lim H, Lee C, Chizen D, Harris G, Hale G, Burger H, Baerwald A. Associations Between Antral Ovarian Follicle Dynamics and Hormone Production Throughout the Menstrual Cycle as Women Age. J Clin Endocrinol Metab. 2015 Dec;100(12):4553-62. doi: 10.1210/jc.2015-2643. Epub 2015 Oct 14. PMID 26465392